CLINICAL TRIAL: NCT01469897
Title: Cost of Care for Juvenile Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrew Zeft, Director, Center for Pediatric Rheumatology, The Cleveland Clinic
Other Study IDs: CCF 11-291
Record Dates: First submitted 2011-11-03; First posted 2011-11-10 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA; Juvenile Idiopathic Arthritis; Cost of Care; Quality of Life; QOL
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project seeks to collect data on healthcare utilization and expenditure rates in Juvenile Idiopathic Arthritis (JIA) patients from across the US, correlate these costs with disease activity and outcome measures and determine methods by which to reduce the economic impact while improving outcomes.

DETAILED DESCRIPTION:
SPECIFIC AIMS AND OBJECTIVES

The specific aims of this registry protocol are:

* To create and maintain a secure online database of patients with JIA
* To collect data elements related to cost of care in patients with JIA
* Compare standard outcome and disease activity measures to health care expenditures in JIA
* To determine methods by which to reduce costs while improving outcomes and quality of care

The study plans to enroll 300 or more subjects from 3 medical centers in the US over a 24 month period. Subjects in the study are patients with Juvenile Idiopathic Arthritis.

Enrollment into the protocol will include key demographic and clinical data including, medication exposures, disease severity, and function including disease-specific data elements; and estimates of health care service utilization and health care expenditures. Data will be collected once per subject within the context of a standard of care visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with JIA by a pediatric rheumatologist according to published criteria.
* Person providing consent must be able to read English.
* Subject (and/or parent/legal guardian) is able to provide informed consent and willing to comply with study procedures.

Exclusion Criteria:

* Subject/ legal guardian is unwilling to provide consent, cannot read English, or does not meet published criteria for JIA.
* Coexisting rheumatologic disorder
* Diagnosis of fibromyalgia
* Participation in a drug trial in the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents, and young adults with JIA within Cleveland Clinic Health System and at several other participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Direct and indirect costs | 6 months prior to enrollment
  Patient's history will be reviewed for the prior 6 months to enrollment for expenses incurred related to JIA and it's treatment. This will be done through chart review and questionnaires completed by the patient/parent.

SECONDARY OUTCOMES:
Health related quality of life questionnaires | Day 1
  Self reported questionnaires will be completed by parent.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zeft, MD, Principal Investigator — Cleveland Clinic Children's Hospital
Locations (3):
- United States (3):
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - The Cleveland Clinic, Cleveland, Ohio
  - Dell Childrens Medical Center of Central Texas, Austin, Texas